CLINICAL TRIAL: NCT01336751
Title: Lantus® (Insulin Glargine[rDNA Origin] Injection) vs Humalog® Mix 75/25 (75% Insulin Lispro Protamine Suspension and 25% Insulin Lispro Injection) as add-on Therapy in Type 2 Diabetes Patients Failing Sulfonylurea and Glucophage (Metformin) Combination Treatment: a Randomized, Open, Parallel Study
Brief Title: Lantus Versus Humalog Mix as add-on Therapy in Type Diabetes Patients Failing Sulfonylurea and Metformin Combination Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4021
Record Dates: First submitted 2011-04-14; First posted 2011-04-18 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Insulin Lispro

ARMS (2):
- Insulin glargine (Experimental): Lantus (insulin glargine) administered subcutaneously 15 minutes before the evening meal for 24 weeks. The initial dosage was 10 units /day for 7 days. This was followed by titration every 7 days by increasing the dosage until control was established. Insulin dosages were increased according to a subject's glucose values determined by Self-monitoring blood glucose (SMBG).
  The starting dosage of metformin or sulfonylurea was the dosage the subject was taking when randomized. The dosage was to remain unchanged during the course of the study. The administration schedule was left to the discretion of the investigator.
  Interventions: Drug: Insulin glargine
- Lispro mix (Active Comparator): Humalog Mix 75/25 (lispro mix) administered subcutaneously 15 minutes before the evening meal for 24 weeks. The initial dosage was 10 units /day for 7 days. This was followed by titration every 7 days by increasing the dosage until control was established. Insulin dosages were increased according to a subject's glucose values determined by self-monitoring blood glucose (SMBG).
  The starting dosage of metformin or sulfonylurea was the dosage the subject was taking when randomized. The dosage was to remain unchanged during the course of the study. The administration schedule was left to the discretion of the investigator.
  Interventions: Drug: 75% insulin lispro protamine suspension and 25 % insulin lispro injection

INTERVENTIONS:
Drug: Insulin glargine — solution for subcutaneous injection
  Other Names: Lantus
  Arms: Insulin glargine
Drug: 75% insulin lispro protamine suspension and 25 % insulin lispro injection — suspension for subcutaneous injection
  Other Names: Humalog
  Arms: Lispro mix

SUMMARY:
Study Primary Objectives:

To compare glycemic control, as measured by hemoglobin A1c (A1C), between insulin glargine and 75% insulin lispro protamine suspension/25% insulin lispro as add-on therapies in subjects who failed oral combination therapy with sulfonylurea and metformin.

Study Secondary Objectives :

To compare the following measures between subjects receiving insulin glargine or 75% insulin lispro protamine suspension/25% insulin lispro:

* Incidence of hypoglycemia
* Change in weight
* Change in serum lipid profile
* Percentage of subjects achieving A1C levels ≤7%

DETAILED DESCRIPTION:
The planned duration of enrollment is 6 months. The study consists of 2 weeks screening phase and a study period that was planned to be 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have given their signed informed consent.
* Males or females between 18 and 79 years of age.
* Diagnosis of type 2 diabetes mellitus for at least one year.
* Patients must have had continuous oral hypoglycemic treatment for at least three months using dosing of: at least half maximally labeled dose of sulfonylurea + at least 1000 mg metformin daily.
* HBA1C ≥ 8 % and ≤11 %, inclusive, as measured at screening (visit 1).
* Patients must have BMI of > 25 kg/m2 at baseline
* Willingness to accept, and demonstrate ability to inject insulin glargine or 75% insulin lispro protamine suspension and 25% insulin lispro injection therapy.
* Ability and willingness to perform SMBG profiles using a plasma glucose meter at least twice a day.
* Patients must be able to understand and willing to adhere to and be compliant with the study protocol

Exclusion Criteria:

* Patients, who have had stroke, MI, coronary artery bypass graft (CABG), percutaneous transluminal coronary angioplasty (PTCA) or angina pectoris within the last 12 months.
* Patients with congestive heart failure requiring pharmacological treatment.
* Patients on non-selective beta blockers (including ocular).
* Patients with impaired renal function, as shown by but not limited to serum creatinine ≥ 1.5 mg/dl (133μmol/L) for males, or ≥ 1.4 mg/dl (124 μmol/L) for females.
* Patients with acute infections.
* Patients with diagnosis of dementia.
* Treatment with systemic steroids or large doses of inhaled steroids.
* Patients with acute or chronic metabolic acidosis, including diabetic ketoacidosis.
* Patients with planned radiological examinations requiring administration of contrasting agents.
* Clinical evidence of active liver disease, or serum ALT 2.5 times the upper limit of the normal range.
* Patients with history of hypoglycemia unawareness.
* Pregnant or lactating females.
* Failure to use adequate contraception (women of current reproductive potential only).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2001-07; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in hemoglobin A1c (HbA1c) levels at week 24 | 24 weeks

SECONDARY OUTCOMES:
Percentage of Patients Achieving Glycosylated Hemoglobin A1c (HbA1c) values ≤ 7.0% at Week 24 | 24 weeks
Percentage of Patients Achieving Glycosylated Hemoglobin A1c (HbA1c) values ≤ 8.0% at Week 24 | 24 weeks
Change from baseline in fasting plasma glucose (FBG) values at week 24 | 24 weeks
Change from baseline in serum lipid values at week 24 | 24 weeks
Number and severity of hypoglycemic events and time of occurrence of hypoglycemic events | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States